CLINICAL TRIAL: NCT03222284
Title: The Usability, Acceptability, and Perceived Value of the Cornerstones4Care Powered by Glooko App
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Healthcare Innovation Technology Lab (Industry)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00022321
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; type 2 diabetes; type ii diabetes; insulin; mobile applications; Diabetes Mellitus; Diabetes Mellitus, Type 2; smartphone application; health application
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group 1 (Experimental): N=10 Device intervention
  1. Cornerstones4Care Powered by Glooko App Visits Day 1 Day 7 Day 28
  Interventions: Device: Cornerstones4Care Powered by Glooko App
- Group 2 (Experimental): N=20 Device intervention
  1. Cornerstones4Care Powered by Glooko App Visits Day 1 Day 28
  Interventions: Device: Cornerstones4Care Powered by Glooko App

INTERVENTIONS:
Device: Cornerstones4Care Powered by Glooko App — Cornerstones4Care Powered by Glooko App is an iOS or Android smartphone application designed to support diabetes management by offering people with diabetes easily accessible, personalized tools for self-monitoring and education. C4C allows people with diabetes to monitor personal health metrics and blood glucose levels, with the aim to achieve participant behavior changes that may contribute to lower hospitalizations, diabetes-related complications and overall healthcare costs.

SUMMARY:
This is a two-armed mixed methods study of participants (n=30) diagnosed with type 2 diabetes who use a blood glucose meter as part of their treatment regimen. Participants will have either two or three visits at HITLAB during the 28-day study period.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the utility and user experience of a mobile application, called Cornerstones4Care Powered by Glooko App (C4C), for persons diagnosed with diabetes type 2.Subjects will be asked to use the Cornerstones4Care Powered by Glooko App for an approximately 20 minute monitored demonstration session, followed by a 28-day period of daily engagement with the application.The Cornerstones4Care Powered by Glooko App lets users input nutrition, medication, exercise and other daily information to assist in the management of diabetes type 2. It also has the ability to sync with connected devices, such as blood glucose monitors. Additionally, the application offers a library of educational content for users.

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed with type 2 diabetes
2. Live in the New York Metropolitan area
3. Be at least 18 years of age
4. Able to read, write, and speak in English
5. Have an iPhone or Android phone
6. Use a blood glucose meter
7. Regularly take insulin by injection
8. Be willing to follow study requirements for a 28-day period

Exclusion Criteria:

1. Not be diagnosed with type 2 diabetes
2. Not living in the New York Metropolitan area
3. Be less than 18 years of age
4. Be unable to read, write, and speak in English
5. Not have an iPhone or Android phone
6. Not use a blood glucose meter
7. Not regularly take insulin by injection
8. Be unwilling to follow study requirements for a 28-day period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-17 (Actual); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
Usage of the Cornerstones4Care Powered by Glooko App as assessed by self-report | 28 days
Device usability as assessed by the System Usability Scale (SUS) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Stan Kachnowski, PhD, MPP, Principal Investigator — Healthcare Innovation Technology Lab
Locations (1):
- Healthcare Innovation and Technology Lab, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No